CLINICAL TRIAL: NCT05907655
Title: Discovering the Functional Role of the Glymphatic System in the Genesis of the Migraine Attack
Brief Title: Study of the Glymphatic System in Migraine
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Roberta Messina, Principal Investigator, IRCCS San Raffaele
Other Study IDs: GR-2021-12374851
Record Dates: First submitted 2023-05-16; First posted 2023-06-18 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Migraine
Keywords: migraine; MRI; glymphatic system; sleep; neuropeptides
MeSH Terms: conditions — Migraine Disorders | interventions — Nitroglycerin; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adult patients with migraine: Diagnosis of migraine, by the ICHD-3 criteria. Age between 18 and 60 years. Female and males. Right-handed
  Interventions: Drug: Nitroglycerin 0.3 MG; Diagnostic Test: MRI; Diagnostic Test: Blood sampling; Device: Sleep profiler
- Healthy controls: Age between 18 and 60 years. Female and males. Right-handed
  Interventions: Drug: Nitroglycerin 0.3 MG; Diagnostic Test: MRI; Diagnostic Test: Blood sampling; Device: Sleep profiler

INTERVENTIONS:
Drug: Nitroglycerin 0.3 MG — Sublingual nitroglycerin will be used to provoke spontaneous-like migraine attacks in migraine patients. A dose of 0.9 mg of sublingual nitroglycerin will be used. The same dose will be administrated to controls.
Diagnostic Test: MRI — The following brain MRI sequences will be acquired before and after nitroglycerin administration: fluid attenuated inversion recovery (FLAIR), 3D T1-weighted inversion recovery prepared gradient echo, diffusion weighted sequence and 3D susceptibility weighted images.
Diagnostic Test: Blood sampling — Plasma levels of neuropeptides involed in migraine will be measured using commercially available enzyme-linked immune-sorbent assay (ELISA) kits. All ELISA will be performed by the same experienced technician who will be blinded for the clinical diagnosis.
Device: Sleep profiler — Sleep architecture will be investigated using the Sleep Profiler. Sleep Profiler is medical device with CE mark which is produced by Advanced Brain Monitoring and distributed throughout Italy exclusively by Medigas. Sleep staging will be automatically performed for 30-second epochs throughout a dedicated software and a standardized and validated procedure. Frontopolar EEG signal waveforms will be visually inspected to confirm the accuracy of the auto-staging.

SUMMARY:
This study aimed to investigate the role of the glymphatic system in the initiation of migraine attacks, using non-invasive magnetic resonance imaging techniques and a validated model of migraine induction by nitroglycerin administration. Secondarily, the relationship between the function of the glymphatic system during nitroglycerin-induced migraine attacks and sleep architecture and plasma levels of migraine-involved neuropeptides will be investigated.

ELIGIBILITY:
Inclusion Criteria:

For patients:

• Diagnosis of migraine, by the ICHD-3 criteria;

For both patients and healthy controls:

* Age between 18 and 60 years;
* Willing and able to comply with scheduled visits.

Exclusion criteria

For patients:

* Overuse of acute medications for headache;
* Continuous or daily headache;
* Other primary headache disorders, with the exception of infrequent tension-type headache.

For healthy controls:

• Any subject with frequent tension type headache, migraine, cluster headache, other pain syndromes or neurological conditions.

For both patients and healthy controls:

* Allergy to nitroglycerin;
* Major psychiatric disorders such as bipolar affective disorder and schizophrenia;
* Cardiovascular diseases that contraindicated the use of nitroglycerin;
* Intracranial hypertension;
* Cerebral haemorrhage;
* Cerebral trauma;
* Pulmonary toxic oedema;
* Closed angle glaucoma;
* Anaemia;
* Pregnancy and breastfeeding;
* Aortic stenosis or significant hypotension (SBP<90mmHg or <100mmHg and symptomatic) precluding nitroglycerin administration;
* Use of sildenafil;
* Any person unable to lie still within the environment of the MRI scanner for the required period to perform the study;
* Any person where MRI scanning is contraindicated (metal implants, pacemaker, claustrophobia, etc.);
* Use of illicit drugs;
* MRI head showing any brain pathology, such as space-occupying lesions;
* Any person unable to understand and follow the instructions of the investigators.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with a diagnosis of episodic migraine without aura, by the standard ICHD diagnostic criteria, will be prospectively recruited. Patients will be allowed to take only one migraine preventive treatment at a stable dose during the study. Healthy controls suffering from any headaches with the exception of infrequent tension-type headache will be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline glymphatic function after nitroglycerin administration | Up to 8 hours
  The DTI-ALPS index will be quantified before and after nitroglycerin administration as an indirect measure of the glymphatic function

SECONDARY OUTCOMES:
Change from baseline plasma levels of neuropeptides after nitroglycerin administration | Up to 8 hours
  ELISA kits will be used to measure the plasma level of neuropeptides involved in migraine pathophysiology before and after nitroglycerin administration
Change from baseline sleep architecture after nitroglycerin administration | Up to 8 hours
  Sleep Architecture will be studied through the Sleep Profiler before and after nitroglycerin administration

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Messina, MD, PhD, Principal Investigator — IRCCS San Raffaele Hospital
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Italy